CLINICAL TRIAL: NCT00639548
Title: Auditory Event-Related Potentials, BIS-Index and Entropy for the Discrimination of Different Levels of Sedation in the ICU Patients
Brief Title: ERPS, BIS and Entropy for Neuromonitoring in ICU Patients
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Haenggi Matthias, Department of Intensive Care Medicine - Inselspital
Other Study IDs: KIM-NMP4
Record Dates: First submitted 2008-03-12; First posted 2008-03-20 (Estimated); Last update posted 2008-03-20 (Estimated); Status verified 2008-03

CONDITIONS: Deep Sedation; Electroencephalography; Event-Related Potentials; Evoked Potentials, Auditory
Keywords: Deep Sedation; EEG; Event-Related Potentials; Evoked potentials, auditory; BIS-Index; Entropy; ICU

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Most critically ill patients receive sedative and analgesic drugs to attenuate discomfort and pain. The excessive use of sedatives and analgesics has undesirable effects for patients. Whereas undersedation is mostly easy to identify, oversedation with its associated problems is more difficult to recognize. Stopping sedation daily helps to avoid gross oversedation, but this is not always possible. Monitoring the depth of sedation is difficult and is currently based on clinical assessment and the use of clinical scoring systems. These scoring systems cannot be applied continuously, they are subjective and the level of consciousness can be altered when sedation is assessed.

Several methods based on the electroencephalogram have been tested to avoid these problems, but the results have been disappointing so far, so the BIS Monitor an dthe Entropy monitor.We have previously shown that the time-locked cortical response to standard external stimuli (long-latency auditory evoked potentials or event-related potentials; ERPs) can discriminate between clinically relevant light to moderate and deep sedation levels in healthy volunteers, when sedation is induced with a combination of propofol or midazolam with remifentanil.

We therefore hypothesized that ERPs may be used to monitor the depth of sedation in ICU patients as well. As the first step to test this hypothesis, we evaluated the use of ERPs to assess the level of sedation in patients undergoing elective major surgery and admitted to the ICU for short term postoperative mechanical ventilation.

DETAILED DESCRIPTION:
Most critically ill patients receive sedative and analgesic drugs to attenuate discomfort and pain. The excessive use of sedatives and analgesics prolongs time on mechanical ventilation, the incidence of nosocomial pneumonia, time spent in the intensive care unit, and increases costs. Strategies to reduce the use of sedatives and analgesics may improve the outcome. Whereas undersedation is mostly easy to identify, oversedation with its associated problems is more difficult to recognize, but should be avoided. While stopping sedation daily helps to avoid gross oversedation, this is not always possible, e.g. due to unstable condition of the patient. Also, accumulation of sedatives and analgesics may occur rapidly, especially in patients with renal and/or liver dysfunction. Monitoring the depth of sedation is difficult and is currently based on clinical assessment and the use of clinical scoring systems. These scoring systems cannot be applied continuously, they are subjective and the level of consciousness can be altered when sedation is assessed.

Several methods based on the electroencephalogram have been tested to avoid these problems, but the results have been disappointing so far. A relatively new method of processed EEG is Entropy®. Entropy is a non-linear statistic parameter which describes the order of random repetitive signals. In patients it translates the anesthesia-induced "calmer", more synchronized EEG into a single parameter. Spectral entropy can reproducibly indicate the hypnotic effects of propofol, thiopental and different anesthetic gases. The most popular method of processed EEG for assessment of sedation is the bispectral index (BIS-Index®). While BIS has been tested and validated for the use in the operation room with different anesthetics, data on its use in the ICU setting at less deep levels of sedation are controversial. The multiple concomitant medications and heterogeneity of underlying pathologies present a further challenge to the use of neuromonitoring in the ICU.

We have previously shown that the time-locked cortical response to standard external stimuli (long-latency auditory evoked potentials or event-related potentials; ERPs) can discriminate between clinically relevant light to moderate and deep sedation levels in healthy volunteers, when sedation is induced with a combination of propofol or midazolam with remifentanil.

We therefore hypothesized that ERPs may be used to monitor the depth of sedation in ICU patients as well. As the first step to test this hypothesis, we evaluated the use of ERPs to assess the level of sedation in patients undergoing elective major surgery and admitted to the ICU for short term postoperative mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years or older

Exclusion Criteria:

* ASA class III or higher history of adverse events during former surgery or anesthesia, neurological impairment in the medical history hearing abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients required an elective thoracic surgical intervention under general anesthesia and who were scheduled to the ICU for postoperative care
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2004-11; Primary Completion 2006-07 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Event related Potentials (Amplitudes, latencies) at different clinically relevant sedation levels | postoperative awakening

SECONDARY OUTCOMES:
BIS-Index at different clinically relevant sedation levels | postoperative awaakening
Entropy at different clinically relevant sedation levels | postoperative awakening

CONTACTS AND LOCATIONS:
Locations (1):
- Departement of Intensive Care Medicine - University Hospital Bern - Inselspital, Bern, Switzerland

REFERENCES:
- [Background] Haenggi M, Ypparila H, Hauser K, Caviezel C, Korhonen I, Takala J, Jakob SM. The effects of dexmedetomidine/remifentanil and midazolam/remifentanil on auditory-evoked potentials and electroencephalogram at light-to-moderate sedation levels in healthy subjects. Anesth Analg. 2006 Nov;103(5):1163-9. doi: 10.1213/01.ane.0000237394.21087.85. PMID 17056949
- [Background] Haenggi M, Ypparila H, Takala J, Korhonen I, Luginbuhl M, Petersen-Felix S, Jakob SM. Measuring depth of sedation with auditory evoked potentials during controlled infusion of propofol and remifentanil in healthy volunteers. Anesth Analg. 2004 Dec;99(6):1728-1736. doi: 10.1213/01.ANE.0000135634.46493.0A. PMID 15562062